CLINICAL TRIAL: NCT02605161
Title: Imaging Blood Brain Imaging Dysfunction in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20150770-01H
Record Dates: First submitted 2015-11-03; First posted 2015-11-16 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Parkinson's Disease; Movement Disorders
Keywords: Blood brain barrier; movement disorder; deep brain stimulation; essential tremor; cervical dystonia; magnetic resonance imaging; neostriatum
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Essential Tremor; Torticollis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease group: * patients diagnosed with Parkinson's disease by a movement disorder specialist from the deep brain stimulation program at The Ottawa Hospital, Civic Campus
  * to undergo pre-operative MRI with contrast
- Control group: * patients diagnosed with either essential tremor or cervical dystonia by a movement disorder specialist from the deep brain stimulation program at The Ottawa Hospital, Civic Campus
  * to undergo pre-operative MRI with contrast

SUMMARY:
The purpose of this study is to evaluate the blood brain barrier in the striatum of patients that have other types of movement disorders compared to patients with Parkinson's Disease that are receiving similar treatment, to determine if a there is a disruption of the blood brain barrier in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the most common neurodegenerative movement disorder of aging. Its cause is unknown. Current evidence supports a stress-diathesis model of pathogenesis whereby some yet-to-be identified environmental trigger conspires with a permissive genetic background to initiate the disease process. Based on neuropathological observations in other neurodegenerative diseases, such as chronic traumatic encephalopathy where pathological protein aggregates form in close association with damaged blood vessels, investigators have hypothesized that the environmental trigger resides in the bloodstream. As a corollary of this hypothesis, investigators propose that the PD pathological process begins in the brain of affected individuals only after disruption of the blood brain barrier (BBB), thereby allowing access of the inciting agent to nigrostriatal axon terminals in the neostriatum. This forms the foundation for the investigators' hypothesis that the BBB in the neostriatum of PD patients is disrupted. Indeed, in a post-mortem study, investigators demonstrated histopathological evidence for significant striatal BBB disruption in sections of striatum from PD subjects relative to age-matched controls. Critics of this study indicate that post-mortem effects may result in artefactual disruption of the BBB, calling into question the validity and relevance of this potentially important finding to PD pathogenesis and progression. Therefore, investigators are performing this imaging study of live PD patients as a follow-up of their convincing post-mortem study to definitively establish whether BBB dysfunction is a feature of PD.

The neostriatal BBB is dysfunctional in PD patients relative to controls and this can be demonstrated by significantly increased parenchymal enhancement on magnetic resonance imaging (MRI).

The results of these studies could have important implications for the understanding of PD pathogenesis. There is emerging evidence that the key pathogenetic event in PD pathogenesis, aggregation of alpha-synuclein, begins within the axon terminals of neurons. The neurons most severely affected in PD reside in the substantia nigra and project to the neostriatum. Demonstrating disruption of the BBB in the PD striatum would render nigrostriatal axon terminals susceptible to a blood-borne disease trigger and allow researchers to generate hypotheses regarding the identity of this trigger. Immune/inflammatory candidates are particularly attractive in this regard. The results this study may also have therapeutic implications. For example, if alpha-synuclein disaggregating agents achieve therapeutic utility in the coming years, our studies may indicate that such agents may be capable of accessing nigrostriatal axon terminals without requiring pharmaceutical or mechanical disruption of the BBB.

ELIGIBILITY:
Inclusion Criteria:

* Disease burden is dominated by motor symptoms such as rigidity, bradykinesia, akinesia, and tremor;
* Medications have been optimized by a movement disorder neurologist;
* Adequate social support to assist with preoperative recovery and problems during subsequent programming;
* No major mood disorder and any mood disorders are medically optimized;
* No major cognitive impairment;
* No underlying medical conditions that would preclude surgery;
* Adequate response to levodopa, as assessed by UPDRS-3 on and off levodopa. All participants has at least a 30% improvement;
* eGRF>30

Exclusion Criteria:

* Disease burden is not dominated by motor symptoms such as rigidity, bradykinesia, akinesia, and tremor;
* Medications have not bee optimized by a movement disorder neurologist;
* There is not adequate social support to assist with pre-operative recovery or problems during subsequent programming;
* Presence of major mood disorders or any mood disorders not medically optimized;
* Presence of major cognitive impairment;
* Presence of underlying medical conditions that would preclude surgery;
* Inadequate response to levodopa;
* eGFR<30

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having movement disorders undergoing deep brain stimulation (DBS) of the internal segment of the globus pallidus for treatment of motor symptoms refractory to medical therapy at the Ottawa Hospital, Civic Campus, will be recruited to participate in this pilot study. The cohort will include 10 PD patients and 10 control subjects. The PD subjects will have received a diagnosis of PD using established clinical criteria following clinical assessment at the Movement Disorders Clinic of The Ottawa Hospital. The 10 control subjects will consist of those undergoing DBS and assessed in the same clinic with a clinical diagnosis of either essential tremor or cervical dystonia.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Degree of contrast enhancement | one year
  Pre-contrast images will be used as mask images and will be digitally substracted from post-contrast images to obtain the "difference" images. From the "difference images", two neuroradiologists blinded to the clinical status of the patient will assess the degree enhancement in the striatum (none,mild, moderate, marked).

SECONDARY OUTCOMES:
Permeability of blood brain barrier in the striatum | one year
  Quantitative assessment of the permeability of the blood brain barrier in the striatum will be assessed using dynamic contrast enhanced MRI. Specifically, the volume transfer constant (Ktrans) will be measured from the striatum in the control and patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh B Nguyen, MD, FRCP, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Warner TT, Schapira AH. Genetic and environmental factors in the cause of Parkinson's disease. Ann Neurol. 2003;53 Suppl 3:S16-23; discussion S23-5. doi: 10.1002/ana.10487. PMID 12666095
- [Background] Gray MT, Woulfe JM. Striatal blood-brain barrier permeability in Parkinson's disease. J Cereb Blood Flow Metab. 2015 May;35(5):747-50. doi: 10.1038/jcbfm.2015.32. Epub 2015 Mar 11. PMID 25757748
- [Background] Schulz-Schaeffer WJ. The synaptic pathology of alpha-synuclein aggregation in dementia with Lewy bodies, Parkinson's disease and Parkinson's disease dementia. Acta Neuropathol. 2010 Aug;120(2):131-43. doi: 10.1007/s00401-010-0711-0. Epub 2010 Jun 20. PMID 20563819
- [Background] Orr CF, Rowe DB, Mizuno Y, Mori H, Halliday GM. A possible role for humoral immunity in the pathogenesis of Parkinson's disease. Brain. 2005 Nov;128(Pt 11):2665-74. doi: 10.1093/brain/awh625. Epub 2005 Oct 11. PMID 16219675